CLINICAL TRIAL: NCT01861145
Title: Intranasal Steroids for the Treatment of Nocturnal Enuresis With Associated Obstructive Sleep Apnea
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to sufficiently enroll or collect follow-up
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Peter Metcalfe, Urologist, University of Alberta
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00032936
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Enuresis; Obstructive Sleep Apnea; Sleep Disordered Breathing
Keywords: Intranasal steroids
MeSH Terms: conditions — Enuresis; Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bed Alarm (Active Comparator): Patients in the control arm will use only the bed alarm for treatment of their enuresis
  Interventions: Device: Bed Alarm
- Bed alarm + intranasal steroids (Experimental): Intervention: Nasonex (Mometasone furoate aqueous nasal spray) Children 5-11: 50 mcg/metered spray, 1 sprays in each nostril daily for 3 months in conjunction with nightly use of the bed alarm.
  Children ≥ 12: 50 mcg/metered spray, 2 sprays in each nostril daily for 3 months in conjunction with nightly use of the bed alarm.
  Interventions: Device: Bed Alarm; Drug: Nasonex

INTERVENTIONS:
Device: Bed Alarm — The bed alarm is a device that is worn at night with a sensor in the child's underwear. The alarm will activate when the child urinates, helping the brain to link the sensation of a full bladder with wakening.
  Other Names: Enuresis Alarm
Drug: Nasonex — Intranasal steroids are used by otolaryngologists as first line treatment for adenotonsillar hypertrophy in children with suspected sleep-disordered breathing and obstructive sleep apnea. The spray helps to shrink the size of the adenoids and tonsils, diminishing the amount of tissue obstructing the child's airway.
  Other Names: Mometasone Furoate Aqueous Nasal Spray
  Arms: Bed alarm + intranasal steroids

SUMMARY:
Enuresis (E) or bedwetting is a common pediatric complaint, and recent research has discovered a link with obstructive sleep apnea (OSA). In children, OSA is often secondary to enlargement of their adenoids or tonsils, and is often successfully treated with a steroid solution given through the nose.

The relationship between SDB and E is incompletely understood. Airway obstruction affects the quality of sleep, as the child will wake as the oxygen levels drop. Abnormal sleep also can decrease the secretion of hormones that affects the kidney's ability to concentrate urine at night, which can result in too much urine in the bladder. Contemporary evidence also suggests that patients with enuresis have abnormal sleep phases, which may impair the communications and inhibition of the bladder.

In previous studies, the investigators have demonstrated that children with E have a high likelihood of having concomitant SDB. The investigators have also demonstrated that children with E and symptoms of SDB do not respond to typical management for bedwetting. Therefore, the investigators propose to treat patients presenting with E with our standard treatments for E (bed alarm) and first line therapy for SDB: Intranasal steroids. This medication helps to decrease the inflammation of the adenoids and tonsils, thereby reducing the airway obstruction. the investigators hypothesize that children with significant symptoms of SDB will improve with the addition of INS, and the investigators hope to see an improvement in their bedwetting, quality of life, and sleep quality as well.

To test this, patents with E will be recruited from the pediatric urology clinic. They will be offered the standard treatment for E, the bed alarm, and the treatment group will be given an intranasal steroid spray. The investigators will then reassess the patients 3 months after treatment, and compare the two groups.

DETAILED DESCRIPTION:
Enuresis (E) is a common pediatric urological complaint. Up to 15% of 5-year old children and 5% of 10-year old children are affected. Despite its prevalence, E is often ineffectively managed. Current treatment modalities include behavior modification, alarm therapy, and pharmacologic treatment. Recently, a significant amount of contemporary research has focused on sleep-disordered breathing (SDB) and its relation to E. This term encompasses a variety of disorders characterized by abnormalities of respiratory pattern or the quantity of ventilation during sleep. Often symptoms of OSA in children may be insidious in nature, and include behavioural problems, hyperactivity, poor school performance, failure to thrive and enuresis.

The relationship between E and OSA has only recently been questioned. Cinar et al. demonstrated 63% complete resolution and 4% partial resolution of E post surgical treatment of upper airway obstruction. Basha et al. had a similar result, with 61.4% of patients having total resolution of NE. The investigators have previously published results on the incidence of SDB in the enuretic population. Using the OSA-18 and PSQ-22 as screening tools for the symptoms of SDB, the investigators found that a significant proportion of patients with enuresis have SDB and the risk is further magnified in patients with abnormal daytime voiding.

The pathophysiology of this relationship is currently under review. With cystometrography, Brooks et al. demonstrated an increase in bladder pressure from 5 to 60 cm H2O with increasing respiratory efforts. Mahler et al. demonstrated that in healthy children exposed to sleep deprivation, disruption in the circadian rhythm resulted in a 68% increase in urine volume, a significant increase in sodium excretion, clearance, and fractional excretion. Sleep deprivation also resulted in higher nighttime blood pressure, and heart rate, which affected sodium regulating hormones, including the renin-angiotension-aldosterone system and ANP. Apneic episodes result in similar fluctuations in sodium excretion, by causing an increase in intrathoracic pressure, increased stretch of the cardiomyocytes, and excretion of atrial and brain natriuretic peptides. Finally, the overall disruption in sleep due to SDB may be the ultimate factor. Healthy children with sleep deprivation demonstrated increased naturiesis, and Yeung et al. demonstration that children with E have abnormal sleep EEG activity with impaired arousability, increased light non-REM sleep, frequent cortical arousals, and impaired wakening.

Enuresis is difficult to treat, and conventional modalities rarely achieve success rates greater than 65%. According to several systematic reviews, enuresis alarms have the highest efficacy rate, and result in an increase in the number of dry nights per week by 4. In a study by Monda et al., 66% of children using enuresis alarms achieved continence by 6 months. Alarms may also reduce treatment failure and relapse that is often associated with the use of medications such as tricyclic antidepressants. Enuresis alarms use a moisture sensor that activates as soon as the child begins to void.

In children, SDB is primarily caused by adenotonsillar hypertrophy, and treatment for OSA begins with a three-month trial of intranasal steroids (INS). INS act by directly reducing adenoidal size by lympholytic action, reducing inflammation, and decreasing the significance of adenoids as a reservoir for infection. In a recent meta-analysis, INS were found to reduce the symptoms of snoring, mouth breathing, and nasal speech by 45-50% when compared to placebo. Similarly, Demirhan et al. showed a mean decrease of adenoid/choana ratio from 86.9% to 56.2% after 8 weeks of fluticasone. In a recent meta-analysis, Zhang et al. found that 5/6 trials showed a significant improvement in nasal obstruction symptoms and reduction in adenoid size with the use of INS.

The investigators' previous data has shown that children with symptoms of SDB and E do not respond to conventional management of E. The investigators therefore propose to trial a novel management approach, by treating the symptoms of SDB with intranasal steroids, in hopes of improving patient's enuresis.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 5-17
* endorse 5/6 questions on the PSQ-22. These questions include: While sleeping, does your child: Ever snore? Snore more than half the time? Always snore? Snore loudly? Have "heavy" or loud breathing? Have trouble breathing, or struggle to breath?
* desire to use the bed alarm

Exclusion Criteria:

* Children <5
* known neurological disorders resulting in neuropathic bowel or bladder disorder including, but not limited to spinal dysraphisms and spinal cord injuries.
* significant congenital bladder anomalies, such as bladder exstrophy or posterior urethral valves
* patients with craniofacial anomalies or syndromes known to be associated with obstructive sleep apnea (i.e. Trisomy 21, muccopolysaccardiosis)

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Degree of improvement in enuresis after a 3 month trial of INS + bed alarm, compared to the bed alarm alone. | 3 months

SECONDARY OUTCOMES:
Changes in OSA-18 and PSQ-22 scores after 3 month trial of INS | 3 months
Adverse effects related to treatments | 3 months
Patient related differences ie obesity, age, sex, and the effect on continence/treatment | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Metcalfe, MD, Principal Investigator — Stollery Children's Hospital and the University of Alberta
Locations (2):
- Canada (2):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Synergy Respiratory Care Centre, Sherwood Park, Alberta